CLINICAL TRIAL: NCT06451211
Title: Phase II Study of Neoadjuvant Immunotherapy Plus Chemotherapy in Borrmann Type 4 and Large Type 3 Gastric Cancer (Neo-ICEBOAT Study)
Brief Title: Neoadjuvant Immunotherapy Plus Chemotherapy in Borrmann Type 4 and Large Type 3 Gastric Cancer
Acronym: Neo-ICEBOAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haibo Qiu, MD, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-FXY-203
Record Dates: First submitted 2024-05-25; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Stomach Neoplasms; Gastric Cancer; Linitis Plastica of Stomach
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab; Oxaliplatin; S 1 (combination); Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab + SOX/XELOX (Experimental): Patients with borrmann type 4 or large type 3 (over 8 cm) gastric cancer, who are deemed to be surgically resectable, are treated with neoadjuvant Tislelizumab (200 mg) and oxaliplatin (150 mg) intravenously on day 1 plus capecitabine (2500 mg) or S-1 (40 mg) orally on day 1-14 in each 21-day cycle. Radical gastrectomy will be performed after 6 cycles, followed by adjuvant chemotherapy (capecitabine or S-1).
  Interventions: Drug: Tislelizumab; Drug: Oxaliplatin; Drug: S-1; Drug: Capecitabine

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200 mg will be administered systemically on day 1 of each cycle in all participants
Drug: Oxaliplatin — Oxaliplatin 150 mg will be administered systemically on day 1 of each cycle in all participants
Drug: S-1 — S-1 40 mg will be administered orally on day 1-14 of each cycle in all participants
Drug: Capecitabine — Capecitabine 2500 mg will be administered orally on day 1-14 of each cycle in all participants

SUMMARY:
The aim of this study is to test the efficacy and safety of immunotherapy plus chemotherapy on people with a relatively rare type of gastric cancer. Participants will take the anti-PD-1 inhibitor (Tislelizumab) and platinum-based chemotherapy (oxaliplatin + capecitabine or oxaliplatin + S-1) in a 3-week cycle, followed by a radical operation after 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed gastric adenocarcinoma,cT1-2N+M0 or cT3-4NanyM0;
* Males or females, aged 18-70 years;
* Gastroscopy and abdominal computed tomography (CT) scan-confirmed typical scirrhous gastric cancer (borrmann type 4) or large type 3 (over 8 cm);
* No peritoneal metastasis confirmed by laparoscopic exploration and with cytological examination of peritoneal washing of the Douglas pouch;
* ECOG performance status 0 or 1;
* Sufficient organ function:

  * white blood cell count > 4*10^9/L, neutrophil cell count > 1.5*10^9/L, hemoglobin > 90 g/L, platelet count > 100*10^9 /L
  * Serum bilirubin ≤ 1.5×upper limit of normal (ULN), AST, ALT ≤ 2.5×ULN
  * Creatinine ≤ 1.5 ×ULN or serum clearance > 60 ml/min
  * INR and aPTT ≤ 1.5 × ULN, only for subjects not receiving anticoagulant therapy;Subjects undergoing coagulation therapy should use a stable dose
* No prior anti-tumor therapy;
* Have signed informed consent before the beginning of treatment.

Exclusion Criteria:

* History of another malignancy within the last five years;
* Previous cytotoxic chemotherapy, radiotherapy or immunotherapy
* Unable to take drugs orally
* Allergic to to any drug of the study regimen;
* Women who are pregnant or breastfeeding or may be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
MPR | up to 2 years
  Major pathologic response, defined as less than 10% residual tumor following neoadjuvant therapy

SECONDARY OUTCOMES:
Adverse Events | up to 2 years
Incidence of surgical complications | up to 2 years
Rate of R0 resection | up to 2 years
OS | up to 5 years
  3-year overal survival
DFS | up to 5 years
  3-year disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, MD, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China